CLINICAL TRIAL: NCT04249349
Title: Preliminary Biomechanical and Usability Study of an Active Ankle-Foot Orthesis for Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0003
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Ankle foot orthosis; Gait; Active orthosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted Gait (Experimental): Participants will receive assisted gait with a motorized ankle foot orthosis. Patient´s gait will be analyzed by a photogrammetry system during device assistance. Session will involve 1 hour of supervised training.
  Interventions: Device: Assisted gait with a motorized ankle foot orthosis

INTERVENTIONS:
Device: Assisted gait with a motorized ankle foot orthosis — The motorized ankle foot orthosis is a powered lower extremity assistance device with an actuated ankle joint. A novel control software has been design and implemented in this device, which allows precise joint movement and recording of data from training session.

SUMMARY:
This research will present the biomechanical assessment of a robotic device for ankle assistance during gait on stroke's survivors with hemiparesis. Gait pattern through an optoelectronic motion capture system will be analyzed. Additionally, ergonomic and comfort aspects will be measured by an adapted spanish version of Quebec User Evaluation of Satisfaction with assistive Technology (QUEST)

DETAILED DESCRIPTION:
This research will present the biomechanical assessment of a robotic device for ankle assistance during gait on stroke's survivors with hemiparesis.

The device is composed by a passive orthosis structure which allows one degree of freedom (DOF) among the sagittal plane and it includes two servomotors attached to the user's foot through velcro strips.

Gait pattern through an optoelectronic motion capture system will be analyzed. Additionally, ergonomic and comfort aspects will be measured by an adapted spanish version of Quebec User Evaluation of Satisfaction with assistive Technology (QUEST)

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis caused by a stroke.
* Age between 18 and 65 years old.
* Post-stroke time more than 6 months.
* Independent walking.
* Minimum 90 degrees of dorsiflexion.
* Muscle tone in plantar flexors less than of equal to 3 on the Modified Ashworth scale.
* Ability to follow instructions.
* Voluntary participation.

Exclusion Criteria:

* Skin alterations in the lower limb.
* Peripherical vascular alterations.
* Alterations in sensitivity in the lower limb.
* Pain of musculoskeletal origin in lower extremities or spine.
* History of frequent falls.
* Cancer
* Previous history or suspected seizures.
* Patient who does not sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Gait Deviation Index without assistance | Baseline
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.
Gait Deviation Index assisted by motorized ankle foot orthosis | Day 1
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.
Patient satisfaction with device: Quebec User Evaluation of Satisfaction with Assistive Technology | Day 1
  Measured with QUEST scale. The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components, Device and Services. Scores of 1 indicate dissatisfaction and scores of 5 indicate high satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pennycott A, Wyss D, Vallery H, Klamroth-Marganska V, Riener R. Towards more effective robotic gait training for stroke rehabilitation: a review. J Neuroeng Rehabil. 2012 Sep 7;9:65. doi: 10.1186/1743-0003-9-65. PMID 22953989
- [Background] Nadeau S, Duclos C, Bouyer L, Richards CL. Guiding task-oriented gait training after stroke or spinal cord injury by means of a biomechanical gait analysis. Prog Brain Res. 2011;192:161-80. doi: 10.1016/B978-0-444-53355-5.00011-7. PMID 21763525
- [Background] Belagaje SR. Stroke Rehabilitation. Continuum (Minneap Minn). 2017 Feb;23(1, Cerebrovascular Disease):238-253. doi: 10.1212/CON.0000000000000423. PMID 28157752
- [Background] Shi B, Chen X, Yue Z, Yin S, Weng Q, Zhang X, Wang J, Wen W. Wearable Ankle Robots in Post-stroke Rehabilitation of Gait: A Systematic Review. Front Neurorobot. 2019 Aug 13;13:63. doi: 10.3389/fnbot.2019.00063. eCollection 2019. PMID 31456681
- [Background] Young AJ, Ferris DP. State of the Art and Future Directions for Lower Limb Robotic Exoskeletons. IEEE Trans Neural Syst Rehabil Eng. 2017 Feb;25(2):171-182. doi: 10.1109/TNSRE.2016.2521160. Epub 2016 Jan 27. PMID 26829794